CLINICAL TRIAL: NCT05358795
Title: Family Connections Cluster RCT in Zambia: Impact of a Youth and Caregiver Intervention on HIV Management Among HIV-positive Youth (Ages 15-21)
Brief Title: Family Connections Cluster RCT in Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: FHI 360 (Other); Arthur Davison Children's Hospital (Other); Tropical Diseases Research Centre (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00020325
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: HIV; Adolescent Development; Adolescent Behavior; Caregivers; Africa
Keywords: HIV; Adolescents; Youth; Caregivers; Africa; Intervention
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Connections Intervention Arm (Experimental): The intervention group sessions aim to 1) improve understanding of HIV among AYA and caregivers; 2) help AYA develop strategies for healthy living (e.g. ART adherence); 3) build AYA capacity to make informed decisions about their sexual and reproductive health; 4) build the capacity of caregivers to support AYA; and 5) help AYA develop life skills to communicate their HIV diagnosis effectively and to plan for their futures. Participants attend group sessions, with caregivers and AYA typically separated for sessions and then brought together sometimes during and sometimes at the end of the sessions, to share information and skills learned. The in-person group intervention will be held twice per month over a period of an estimated 6 months for a total of 10 sessions. Trained facilitators will deliver the intervention at the clinics. Health clinic staff will be available as technical experts to answer clinical questions.
  Interventions: Behavioral: Family Connections
- Standard of Care Comparison (No Intervention): The control group will receive the standard of care during the study for AYA living with HIV in these public health care facilities and communities. The 20 facilities included in the research have been trained to operate under the standard protocols endorsed by the Zambia Ministry of Health. There can be variations in how these standards are adhered to and if special programming is provided for youth, such as youth group meetings and special youth clinic hours. Standard of care services per the 2020 Zambia Consolidated Guidelines include routine clinical care for HIV treatment including laboratory testing (CD4, VL tests); adherence counseling, with enhanced adherence counseling for clients with unsuppressed viral loads; multi-month dispensing of ART including differentiated service delivery for stable clients; screening and treatment of sexually transmitted infections (STIs); prevention and screening for opportunistic infections; and clinical monitoring of kidney and liver function.

INTERVENTIONS:
Behavioral: Family Connections — Family Connections is based on the WHO endorsed Positive Connections manual.
  Arms: Family Connections Intervention Arm

SUMMARY:
This study will evaluate the impact of Family Connections, a family-based group intervention for adolescents and young adults (AYA) living with HIV and their family caregivers, on achieving HIV self-management defined as having an undetectable viral load (VL) and low self-stigma (a score of 1 or less), among older adolescents and young adults (AYA) ages 15-to-21 years. The intervention seeks to increase social and family support and decrease self-stigma among AYA, so they may improve their medication adherence and achieve an undetectable viral load. Findings will fill a critical gap in available evidence-based intervention options for improving the HIV-related outcomes and wellbeing of HIV-positive AYA in sub-Saharan Africa.

DETAILED DESCRIPTION:
BACKGROUND/INTRODUCTION

A dearth of programs exist that actively promote HIV self-management among older adolescents and young adults (AYA) in sub-Saharan Africa (SSA). Literature on chronic illness has identified the following skills for promoting self-management: problem-solving, decision-making, resource utilization, formation of a patient-provider partnership, action planning, and self-tailoring skills to one's own situation. While there is an international call to support HIV self-management among adolescents, the reality is that AYAs living with HIV in SSA often do not have access to youth-specific services or opportunities to build life skills. Some clinics hold monthly AYA peer group meetings, however such meetings are typically vulnerable to changes in staff and funding; are often not systematically incorporated into service provision; and do not involve AYAs' family members.

There is also lack evidence on how HIV self-management differs by AYAs' developmental characteristics. Adolescence is a period characterized by intense physical, cognitive, and emotional growth and a desire for independence. Furthermore, data show that some youth living with HIV experience delayed cognitive development, particularly youth that are perinatally infected with HIV. Despite these data, studies rarely examine program impact accounting for variations in AYAs' development. Furthermore, evidence exists that managing chronic illnesses has negative impacts on caregivers and families, particularly in low-income and highly stigmatized environments.

Peer group interventions, however, show promise in reducing HIV-related stigma in SSA among adults and in supporting adolescent ART adherence. Given that HIV is a highly stigmatized chronic illness, peer groups provide a safe environment in which to share experiences and learn from others who understand the day-to-day reality of living with HIV. There is also a growing body of literature from SSA, including Zambia, calling for interventions to involve families in supporting AYA living with HIV to self-manage HIV and to promote family involvement as AYA transition into adulthood and adult HIV services. While experts agree on the need for family-centered approaches and peer support groups, few family-based interventions exist that specifically address the needs of older AYAs aged 15-21 years.

In response to the lack of interventions to promote HIV self-management among AYA that harness the support of caregivers, the study team developed Family Connections- a family group-based intervention. In the study team's earlier pilot study of Family Connections the team adapted an existing adolescent support group guide called Positive Connections (The United States President's Plan for AIDS Relief using mixed-methods formative research. The study team also updated the AYA support group materials and developed a corresponding support group component for caregivers. The feasibility and acceptability of Family Connections was tested in an randomized controlled trial (RCT) among older adolescents (15 to 19 years) and their caregivers in two clinics in Ndola, Zambia. Fifty adolescent/caregiver pairs (100 individuals) were enrolled. Study results found that Family Connections was highly feasible and acceptable. Of the 24 adolescent/caregiver pairs assigned to the intervention arm, 88% attended eight or more of the 10 Family Connections sessions together, and most adolescents (96%) and all caregivers would recommend the intervention to their peers. Although not powered to find differences in outcomes, the prior pilot study showed a signal for efficacy in reducing adolescents' HIV-related feelings of worthlessness (I: 54% to 22% vs. C:38% to 35%, p=0.06) and shame (I: 58% to 30% vs. C:54% to 58%, p=0.07), and reducing caregiver burden (mean scores: I: 0.16 to -0.25 vs. C: -0.15 to -0.25, p=0.08).

Building off this pilot study, this cluster randomized controlled trial (CRCT) will contribute to the field of HIV empirical research and care practices by testing the impact of a feasible and acceptable family-based intervention on increasing the proportion of 15- to 21-year-old AYA who achieve HIV self-management defined as having an undetectable viral load and low self-stigma. This study will also help improve the understanding of how cognitive and developmental processes may moderate intervention outcomes among AYA.

STUDY AIMS:

The specific aims of the research are to:

Aim 1: Assess the impact of Family Connections on achieving HIV self-management defined as having an undetectable viral load (VL <20 copies/mL) and low self-stigma, among AYA. A cluster randomized controlled trial will be conducted comparing 200 pairs of AYA and caregivers at 10 intervention health facilities versus 200 pairs at 10 control health facilities (n=800 total: 400 AYA, 400 caregivers).

Aim 2: Assess the impact of Family Connections on caregiver burden (e.g., How often does the caregiver feel stressed between caring for adolescent and trying to meet other responsibilities for family or work?) and social support among the 200 AYA caregiver participants in the intervention arm versus the 200 AYA caregiver participants in the control arm (n=400).

Aim 3: Examine if the impact of Family Connections on AYAs' HIV self-management is moderated by developmental differences among youth assessed through measures of cognitive functioning, executive functioning, impulse control, and emotional regulation.

STUDY DESIGN

This study is a multi-site, pair-matched CRCT to evaluate the impact of the Family Connections intervention on achieving undetectable VL among AYA living with HIV. The study team will enroll pairs of AYA living with HIV (ages 15-21) and their caregivers in 20 matched pairs of HIV clinics in Copperbelt Province. The team will enroll and collect baseline data, including a VL test, from an estimated 500 to 700 AYA 15-to-21 years living with HIV in Copperbelt Province and 500 to 700 of their caregivers. The range of participants enrolled is provided as it depends on the proportion of youth initially enrolled who have a detectable VL or high self-stigma at baseline. Based on prior research, approximately 20% of AYA enrolled in the study will have an undetectable viral load. These participants will end study participation at that point. An estimated 35 AYA/caregiver pairs in each clinic will be enrolled until there are approximately 400 AYA participants with a detectable VL or high self-stigma and their caregivers who will continue in the study. After a run-in period, during which study procedures will be refined and facilitators will hold Family Connection sessions, the study will commence in 4 clinics (2-matched pairs) in the Copperbelt Province, and then roll out to the remaining clinics in the Copperbelt. Data collection will occur at baseline, midline (at the end of the Family Connections intervention, approximately six months after baseline), and endline (about six months after midline), and will consist of a survey among caregivers and AYA, a blood draw for AYA, and a point of care (POC) urine adherence test for AYA taking Tenofovir as part of their antiretroviral therapy (ART). The 20 clinics have been pair-matched by number of AYA on ART, and location type. One clinic within each of the matched pairs will be randomly assigned to receive the Family Connections intervention, consisting of 10 in-person group sessions that will take place over an estimated 6 months. The other clinic in the matched pair will be assigned to a standard of care control group. The main comparison will be based on the effect at midline after the 6 months of intervention in the intervention group. Additional contrasts will be tested to examine changes of effects over time (e.g., at endline).

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria for AYA include:

* being between 15 and 21 years,
* HIV positive and aware of their HIV status,
* on ART for at least 6 months,
* on first-line ART,
* living within 30-minutes, by personal transportation, of the clinic by self-report,
* being available to attend 10 sessions over 6 months,
* being available for the next 14 months,
* and speaks one of the study languages, English or Bemba

Eligibility criteria for the caregiver is:

* being 22 years of age or older,
* does not work at the study clinic,
* living within 30-minutes, by personal transportation, of the clinic by self-report,
* caring for an AYA who meets the study eligibility criteria,
* being available to attend 10 sessions over 6 months,
* being available over the next 14 months,
* and speaks one of the study languages English or Bemba.

Being a biological parent or family member is not an eligibility criterion.

Exclusion Criteria:

The only exclusion criteria are not fulfilling the inclusion criteria.

-

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1386 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with undetectable viral load and low self-stigma | ~ 6 months from baseline to midline
  Defined as having <20 RNA copies/mL and scoring 1 or less on a 3 point self-stigma scale among adolescent and youth participants

SECONDARY OUTCOMES:
Number of caregivers experiencing caregiver burden measured using the Zarit Burden Interview | ~ 6 months from baseline to midline
  Zarit Burden Interview adapted 12-item 3 point Likert-scale (0=never, 1=sometimes, 2=Always) with higher scores indicating more challenges/burdens experienced in caregiving (among caregivers)
Number of caregivers with higher social support measured with Medical Outcomes Study Social Support Survey (MOS-SS) | ~ 6 months from baseline to midline
  Medical Outcomes Study Social Support Survey (MOS-SS), 20-items, 5-point Likert Scales (1=none of the time; 2= a little of the time; 3= some of the time; 4=most of the time, 5=all of the time), with higher scores indicating receipt of greater social support (among caregivers)
Number of adolescent and youth participants with cognitive challenges assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) pediatric cognitive function scale | ~ 6 months from baseline to midline
  Patient-Reported Outcomes Measurement Information System (PROMIS) pediatric cognitive function adapted through cognitive interviewing (abbreviated 7-item, 5 point Likert-scales with 5=never; 4= a little of the time; 3= sometimes; 4=most of the time, 5=always), with a higher score assessing more difficulties in cognitive abilities/everyday tasks, in the past 4 weeks.
Number of adolescent and youth participants with emotional regulation challenges measures using the Difficulties in Emotion Regulation Scale (DERS-SF) | ~ 6 months from baseline to midline
  Difficulties in Emotion Regulation Scale (DERS-SF), abbreviated 18-items, 5-point Likert scales (5=never; 4= a little of the time; 3= sometimes; 4=most of the time, 5=always), with a higher score assessing greater difficulties identifying/managing emotions.

CONTACTS AND LOCATIONS:
Overall Officials: Julie A. Denison, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Gershom Chongwe, PhD, Principal Investigator — Tropical Diseases Research Center
Locations (1):
- Copperbelt Province Clinics, Ndola, Copperbelt, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Will deposit data into an existing data repository for future research (explain): After the study is completed, the de-identified, archived data will be transmitted to and stored in a Data Repository determined in consultation with the NIH Program Officer, for use by other researchers including those outside of the study. Permission to transmit data to a Data Repository will be included in the informed consent. Blood samples will not be stored for future research purposes.
Supporting Information: Study Protocol
Time Frame: Once the data is de-identified it may be shared in a repository.
Access Criteria: The team plans to place the data in an open access repository.

REFERENCES:
- [Derived] Schue JL, Mainga T, Nonyane BA, Peterson TL, Miti S, Chongwe G, McCarraher DR, Denison JA. Impact of a youth and caregiver intervention on HIV self-management among youth living with HIV: a protocol for the Family Connections cluster RCT in Zambia. Trials. 2026 Jan 28. doi: 10.1186/s13063-026-09455-3. Online ahead of print. PMID 41606621